CLINICAL TRIAL: NCT05187286
Title: Expanded Access for Apixaban
Status: Available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-826
Record Dates: First submitted 2021-11-16; First posted 2022-01-11 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

MeSH Terms: interventions — apixaban

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Apixaban — Administered as directed by treating physician
  Other Names: Eliquis

SUMMARY:
This is an expanded access designed to provide access to apixaban for eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with Congenital or Acquired Heart Disease Requiring Chronic Anticoagulation for Thromboembolism Prevention
* Previously participated in the CV185-362 study and was on apixaban for 1 year or until treatment was no longer required

Exclusion Criteria:

* Weight less than 5 kg or greater than 35 kg

Other inclusion/exclusion criteria apply

Ages: 28 Days to 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Pre-Approval Access (PAA) Healthcare Practitioner Requests — https://www.bms.com/healthcare-providers/early-patient-access-to-investigational-medicine/investigational-drugs-available.html
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome